CLINICAL TRIAL: NCT05990478
Title: Contrast-Enhanced Mammography With Early and Delayed Acquisitions in the Assessment of the Extent of Residual Disease Following Neoadjuvant Treatment in Patients With Breast Cancer
Brief Title: A Study of Contrast-Enhanced Mammography (CEM) Scans in People With Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Challenges to participant accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-224
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; Memorial Sloan Kettering Cancer Center; 23-224
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Breast Cancer: Participants will have a diagnosis of breast cancer
  Interventions: Diagnostic Test: Contrast-Enhanced Mammography; Diagnostic Test: Breast MRI

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Mammography — Participants will have pre- and post-treatment CEM of the affected breast
  Other Names: CEM
Diagnostic Test: Breast MRI — Pre- and post-NAT breast MRI will be performed for all participants

SUMMARY:
The purpose of this study is to find out whether Contrast-Enhanced Mammography/CEM scans performed 2 minutes and 6 minutes after receiving Iohexol contrast dye can be used to identify the amount of residual disease in the breast following neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any women >18 years of age at time of informed consent
* Diagnosed with breast cancer and schedule for NAT

Exclusion Criteria:

* History of kidney disease, creatinine level >1.3 or eGFR <45.
* Known allergic reaction to gadolinium or iodinated contrast media.
* Contraindication to contrast-enhanced breast MRI.
* Lesion not included in the field of view of either pre- or post-NAT MRI or CEM
* Presence of pacemakers or automated implantable cardioverter defibrilator
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the participant's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Compare the sensitivity and specificity of Contrast-Enhanced Mammography/CEM with standard 'early' acquisition to CEM with delayed acquisition | Up to 1 year
  compare the sensitivity and specificity of CEM with standard 'early' acquisition to CEM with delayed acquisition, in detecting breast cancer lesions with pathological complete response (pCR) after NAT.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Machado Horvat, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org